CLINICAL TRIAL: NCT02197741
Title: The Effect of an Additional Bolus Application in Patients With Intrathecal Opiate Administration - a Pilot Study
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2014-15
Record Dates: First submitted 2014-07-04; First posted 2014-07-23 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Pain Syndrome
MeSH Terms: interventions — Opiate Alkaloids

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- opiate without bolus: continuous opiate administration without bolus application
  Interventions: Drug: opiate with bolus
- opiate with bolus: continuous opiate administration with additional bolus application
  Interventions: Drug: opiate with bolus

INTERVENTIONS:
Drug: opiate with bolus

SUMMARY:
An additional, intermittent bolus application in patients with intrathecal opiate administration for chronic pain syndrome may have a positive effect on the effectiveness of the treatment. Thus, the effect of an additional, intermittent bolus application in patients with intrathecal opiate administration was therefore investigated.

Patients already equipped with an intrathecal opiate pump were enrolled into the study. Each patient was submitted to two treatment periods in randomly chosen order (cross-over design): 1. standard treatment (continuous opiate administration) and 2. continuous opiate administration with intermittent opiate bolus application. Both treatment periods lasted 14 days. Patients were asked to record pain intensity, side effects and satisfaction with the treatment.

The following hypotheses were tested:

* The application of additional opiate boli results in significantly lower pain intensity.
* The application of additional opiate boli does not result in a higher rate of adverse Events.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain syndrome
* intrathecal opiate pump
* signed informed consent

Exclusion Criteria:

* younger than 18 years
* other (than opiate) intrathecal drug administration
* discontent with intrathecal opiate therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals with chronic pain syndrome
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
change in pain intensity | day 0. day 14, day 28
  numeric rating scale from 0 to10

SECONDARY OUTCOMES:
change in satisfaction with treatment outcome | day 0, day 14, day 28
  numeric rating scale from 0 to 10
side effects | from day 0 to day 28
  occurrence rate of side effects

CONTACTS AND LOCATIONS:
Overall Officials: Tim Reck, MD, Principal Investigator — Center for Pain Medicine